CLINICAL TRIAL: NCT03255616
Title: Low Back Pain: Unveiling the Contribution of Motor Control Adaption Using Biomechanical Modeling and Neuroimaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other); Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Michael Meier, Principal Investigator, Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Project_X
Record Dates: First submitted 2017-08-14; First posted 2017-08-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental): Spine kinematics assessment during daily activities and brain responses to thoracolumbar mechanical and vibrotactile stimulation
  Interventions: Other: mechanical stimulation; Other: vibrotactile stimulation
- Low back pain patients (Experimental): Spine kinematics assessment during daily activities and brain responses to thoracolumbar mechanical and vibrotactile stimulation
  Interventions: Other: mechanical stimulation; Other: vibrotactile stimulation

INTERVENTIONS:
Other: mechanical stimulation — mechanical non-painful low- and high pressure stimuli to thoracolumbar segments of healthy subjects and low back pain patients
Other: vibrotactile stimulation — non-painful vibrotactile stimulation within a frequency range between 20-150Hz to thoracolumbar segments of healthy subjects and low back pain patients

SUMMARY:
This project aims to reveal the potential sensorimotor reorganization of sensory input in low back pain patients and its association with different motor control strategies in LBP.

DETAILED DESCRIPTION:
Background: Low back pain (LBP) is a major health issue. Treatment of chronic LBP is still a major challenge due to a lack of pathophysiological understanding. Thus, understanding LBP pathophysiology is a research priority. Adaptions of motor control likely play a significant role in chronic or recurrent LBP because motor control is crucial for spine posture, stability and movement. Different motor adaption strategies exist across individuals with LBP and two phenotypes representing the opposite ends of a spectrum have been suggested; i.e. "tight" control and "loose" control over trunk movement. The former would be associated with reduced trunk motor variability, the later with increased trunk motor variability. This conceptual framework is very useful to explain maintenance and aggravating of LBP because motor control adaptations are expected to have long-term consequences, such as increased spinal tissue loading, associated with degeneration of intervertebral discs and other tissues. Several knowledge gaps need to be addressed to test the validity of this framework: 1) Do loose/tight control phenotypes indeed exist and/or do other motor control adaption strategies exist? 2) Is reduced/altered paraspinal proprioceptive input associated with LBP related to neuroplastic cortical changes, thereby affecting the organizational structure in sensorimotor cortices and top-down trunk motor control? 3) Do psychological factors influence the organizational structure in sensorimotor cortices and motor control strategies? To address these knowledge gaps, the objectives of the current project are: I) To establish motor control phenotypes in LBP. Proprioceptive weighting and biomechanical assessment of dynamic movement tasks, including subject-specific spine kinematic variability and its relationship to pain duration, negative pain-related cognitions, segmental loadings and paraspinal muscle forces, will be performed. II) To test whether cortical proprioceptive maps differ between healthy subjects and patients with LBP. Brain activation in response to thoracolumbar vibrotactile stimulation will be interrogated using functional magnetic resonance imaging data and univariate and multivariate analysis based on machine learning. III) To test whether proprioceptive maps demonstrate a relationship to spine kinematic patterns, pain duration and negative pain-related cognitions in LBP patients.

ELIGIBILITY:
Inclusion criteria healthy subjects:

* Aged between 18 and 60
* Written informed consent after being informed

Inclusion criteria low back pain patients:

* Aged between 18 and 60
* Low back pain for more than 1 week

Exclusion criteria healthy subjects:

* Consumption of alcohol, drugs, analgesics within the last 24 h
* Pregnancy
* acute and/or low recurrent back pain within the last 3 months
* Prior spine surgery
* Other chronic pain condition
* history of psychiatric or neurological disorders
* MR-contraindications
* Body mass index (BMI) > 30 kg/m2

Exclusion criteria low back pain patients:

* Consumption of alcohol, drugs, analgesics within the last 24 h
* Pregnancy
* Specific causes for the back pain (ruled out by the clinician)
* Prior spine surgery
* History of psychiatric or neurological disorders
* MR-contraindications
* Body mass index (BMI) > 30 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent (BOLD) responses | MR assessment, 30 minutes
  supraspinal BOLD responses induced by mechanical and vibrotactile stimulations of the back recorded by means of functional magnetic resonance imaging (fMRI)
Spine kinematics | Spinal kinematics assessment, 120 minutes
  Sagittal and frontal plane lumbar and thoracic spinal curvature angles
Spine biomechanics: muscle forces | Spinal kinematics assessment, 120 minutes
  segmental muscle forces (N/mm) during dynamic tasks
Spine biomechanics: segmental loading | Spinal kinematics assessment, 120 minutes
  segmental loading (N) during dynamic tasks
Proprioceptive repositioning errors | Proprioceptive assessment, 10 minutes
  Sagittal plane repositioning errors assessed through lumbar and thoracic spinal curvature angles
Center of pressure displacements | Postural stability assessment, 20 minutes
  Center of pressure displacements during vibrotactile stimulation while standing on a force plate

SECONDARY OUTCOMES:
Segmental movement | MR assessment, 20 minutes
  Displacement (intervertebral angles) of the stimulated and adjacent spinal segments during mechanical pressure using dynamic T2 scans
Fear of movement | Medical assessment, 5 minutes
  score of the Tampa Scale of Kinesiphobia (TSK) questionnaire
Fear Avoidance Beliefs | Medical assessment, 5 minutes
  scores of the Fear Aovidance Beliefs questionnaire (FABQ) in low back pain patients
Level of disability | Medical assessment, 3 minutes
  scores of the Oswestry Disability Index (ODI) in low back pain patients
Pain characteristics | Medical assessment, 1 minutes
  Pain quality assessment using the PainDETECT questionnaire in low back pain patients
Perception of the back | Medical assessment, 2 minutes
  Assessment of self-perception of the back using the Fremantle Back Awareness Questionnaire
State and Trait anxiety | Medical assessment, 2 minutes
  scores of state and trait anxiety (STAI) questionnaire
Perceived harmfulness of back stressing movements | Medical assessment, 15 minutes
  Assessment of the perceived harmfulness of back stressing movements using the electronic version of the PHODA questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Meier, PhD, Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to share the fMRI dataset in BIDS format on "openfmri.org"